CLINICAL TRIAL: NCT00013260
Title: An Integrated Model of Primary Care in Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MPC 97-010
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Depression
Keywords: Case management; Nurse intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Integrated model of primary care

INTERVENTIONS:
Procedure: Integrated model of primary care

SUMMARY:
Managed care systems rely on primary care providers as gatekeepers to make sensible decisions regarding the use of expensive health care resources. While this model has some intuitive appeal in terms of its potential for decreasing health care costs, it may not be applicable in VA medical centers, where patients are often medically complex and socioeconomically vulnerable. Thus, other strategies to integrate generalist and specialist care are required.

DETAILED DESCRIPTION:
Background:

Managed care systems rely on primary care providers as gatekeepers to make sensible decisions regarding the use of expensive health care resources. While this model has some intuitive appeal in terms of its potential for decreasing health care costs, it may not be applicable in VA medical centers, where patients are often medically complex and socioeconomically vulnerable. Thus, other strategies to integrate generalist and specialist care are required.

Objectives:

Our objective is to evaluate the effectiveness of an integrated model of primary care for veterans with alcohol dependence and/or depression in which mental health clinical nurse specialists (CNS) are placed within the General Medicine Clinic (GMC). Our primary outcomes are patients� disease-specific mental health symptoms (Beck Depression Inventory: BDI) and satisfaction with care (RAND). Secondary outcomes include quality of care, health services utilization, and health care costs.

Methods:

This is a randomized, controlled trial comparing patients in two GMC firms. After physicians in both firms were trained in the diagnosis and brief treatment of the two conditions, the two firms were randomized into one of two conditions. Patients in both firms are screened for depression. Patients who screen positive for depression and give written informed consent are enrolled. In the control firm, depression screening results are provided to the primary care physician. In the integrated primary care firm, results are shared with the primary care provider, along with having a mental health clinical nurse specialist in the GMC who is available to implement and support treatment decisions. Telephone interviews are conducted at three and 12 months after enrollment to collect outcome data by persons blinded to the study hypotheses. Data will also be collected using local VA databases. Data analysis will utilize generalized estimating equations to account for the repeated measures design, clustering of patients within physicians, and clustering of physicians within clinics.

Status:

Data collection was completed during August, 2000. Data analyses for the one-year follow-up results are in process.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of depression (ie, major depression, dysthymia, or partially remitted major depression);
* received primary care from the General Medicine Clinic; and 3) access to a telephone. Patients were excluded if they were: 1) incompetent for interview (eg, active psychosis, dementia documented in medical chart); 2) residents of a nursing home;
* actively suicidal (ie, stated plans/means and/or had suicide attempt during past two years);
* seen in a VA mental health program (made a visit during the previous 30 days and had a future appointment scheduled);
* active cocaine or opiate abusers;
* history of bipolar disorder; or
* terminally ill (ie, death expected with 12 months) using criteria successfully employed in previous studies of veterans in primary care

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Estimated)
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris Weinberger, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, North Carolina, United States